CLINICAL TRIAL: NCT01029392
Title: Prevalence of Vitamin D Deficiency in Type 1 Diabetes Mellitus and Effect on Insulin Requirements After Supplementation With Vitamin D-A Pilot Study
Brief Title: Prevalence of Vitamin D Deficiency in Type 1 Diabetes Mellitus and Effect of Supplementation on Insulin Requirements
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Peter Gerrits, MD, Principal Investigator, Corewell Health East
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2009-189
Record Dates: First submitted 2009-12-09; First posted 2009-12-10 (Estimated); Results first posted 2017-04-17 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2016-12

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Diabetes; Type I; Newly Diagnosis Type I Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Patients with clinically significantly low Vitamin D levels (<30 ng/mL) were supplemented with Vitamin D and compared to patients with normal vitamin D levels (50-80 nG/mL).
Oversight: Data Monitoring Committee: No

ARMS (2):
- Required Vitamin D (Experimental): Those children whose Vitamin D level was low (<30 ng/mL) are given Vitamin D supplementation
  Interventions: Drug: Vitamin D
- Normal Vitamin D (No Intervention): Those children whose Vitamin D level was normal (50-80 ng/mL) did not receive Vitamin D supplementation

INTERVENTIONS:
Drug: Vitamin D — 2000iu once a day
  Other Names: cholecalciferol
  Arms: Required Vitamin D

SUMMARY:
Our objective is to demonstrate that providing supplemental vitamin D to children with new onset DM will significantly decrease the levels of HbA1c and insulin requirement by the following methods.

1. Identify how often vitamin D levels are low in patients with new onset Type 1 diabetes mellitus (DM).
2. Record the hemoglobin A1c (HbA1c) level (which reflects the average blood sugar level over the past few months) and document insulin requirements before and after vitamin supplementation is given.

Hypothesis: Maintaining vitamin D levels >30 ng/ml will decrease HbA1c and insulin requirements.

DETAILED DESCRIPTION:
New onset type 1 DM patients who present at William Beaumont Hospital, Royal Oak or to the Pediatric Endocrine Clinic will be approached about the study at their presentation and time will be given for the patient and family to discuss and ask questions regarding the study. Patients will then be enrolled following informed consent. Glucose levels and insulin requirements will be monitored continuously from the faxed weekly logbooks from the point of diagnosis for 3 months (as standard practice for all newly diagnosed diabetic patients in our clinic). At the baseline visit a Vitamin D level will be drawn and frozen for 3 months prior to processing. .After 3 months vitamin D, calcium, alkaline phosphatase, phosphorus and other standard of care lab draws will be done. Approximately an additional 3 tsp of blood will be taken. All female subjects of child bearing potential will have a pregnancy test done. EMLA cream to anesthetize the area will be used prior to blood draw. A vitamin D level of <30 ng/ml is considered insufficient and the patient will then be given vitamin D supplement. The vitamin D level, calcium, alkaline phosphatase and phosphorus will be rechecked at 6 months (additional 3 tsp of blood) . Glucose levels and insulin requirements will be monitored continuously from the faxed weekly logbooks again for another 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed type I DM.
* Age <18 years

Exclusion Criteria:

* Pregnancy

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Actual)
Dates: Start 2009-11; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Gerrits, MD, Principal Investigator — Corewell Health East
Locations (1):
- WilliamBH, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
No data sharing.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Blood vitamin D level checked to assign to treatment or no-treatment arm
Groups:
- Vitamin D Supplement: Those who had a Vit D level of < 30 ng/mKL
  Vitamin D: 2000 IU once a day
- No Vitamin D Supplementation: Screening vitamin D level in normal range for children (50-80 ng.mL)
Period: Overall Study
Arm/Group | Vitamin D Supplement | No Vitamin D Supplementation
Started | 37 | 38
Completed | 17 | 27
Not Completed | 20 | 11
Not completed — Withdrawal by Subject | 18 | 11
Not completed — Physician Decision | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Those Requiring Vit D Supplement: Those who had a Vit D level of < 30
  Vitamin D: 2000iu once a day
- No Vit D Supplementation: Normal vitamin D levels No Vitamin D supplement
- Total: Total of all reporting groups
Arm/Group | Those Requiring Vit D Supplement | No Vit D Supplementation | Total
Number analyzed (Participants) | 37 | 38 | 75
Age, Categorical [Count of Participants; unit: Participants] — Population: 20 patients in the Vitamin D Supplement arm and 11 patients in the No-Vitamin D supplement arm were withdrawn and not analyzed.
  Participants
    number analyzed (Participants) | 17 | 27 | 44
    <=18 years | 17 | 27 | 44
    Between 18 and 65 years | 0 | 0 | 0
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.4 (4.2) | 8.9 (4.1) | 9.95 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 22 | 23 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 2 | 9
  White | 28 | 31 | 59
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 37 | 38 | 75

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin A1c
Description: Change in hemoglobin A1c calculated as a percentage change from baseline measurement
Time Frame: 6 months
Population: 20 patients in the Vitamin D Supplement arm and 11 patients in the No-Vitamin D supplement arm were withdrawn and not analyzed.
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Groups:
- No Vitamin D Supplementation: Those with normal vitamin D levels (50-80 ng/mL) No vitamin D supplemenation
Arm/Group | Those Requiring Vit D Supplement | No Vitamin D Supplementation
Number analyzed (Participants) | 17 | 27
percentage change from baseline | 2.67 (0.58) | 1.05 (0.58)

2. Secondary Outcome: Change in Insulin Requirements
Description: Percentage change from baseline number of units of lantus insulin over 6 months.
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage change of baseline insulin
Arm/Group | Vitamin D Supplement | No Vitamin D Supplementation
Number analyzed (Participants) | 17 | 27
percentage change of baseline insulin | 2.62 (4.05) | 1.80 (1.55)

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Those Requiring Vit D Supplement: Those who had a Vit D level of < 30 ng/mL Vitamin D: 2000iu once a day
- No Vit D Supplementation: Normal vitamin D levels (50-80 ng/mL) No vitamin D supplementation
Arm/Group | Those Requiring Vit D Supplement | No Vit D Supplementation
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/38
Other Adverse Events (participants affected / at risk) | 0/37 | 0/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Those Requiring Vit D Supplement (N=37) | No Vit D Supplementation (N=38)
Increased dose of Vitamin D needed (Endocrine disorders) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes